CLINICAL TRIAL: NCT02679768
Title: SAFE II: Can Electronic Self-monitoring With Closed Loop Feedback Focusing on Regulation of the Sleep-wake Cycle Reduce Relapse of Depression After Discharge From a Psychiatric Ward?
Brief Title: Electronic Self-monitoring on Regulation of the Sleep-wake Cycle to Reduce Relapse of Depression After Discharge
Acronym: SAFEII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Klaus Martiny, Senior Consultant, Clinical Associate Research Professor, Ph.D., Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAFEII
Record Dates: First submitted 2016-02-08; First posted 2016-02-10 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circadian Reinforcement Therapy (Active Comparator): Circadian reinforcement therapy
  Interventions: Behavioral: Circadian Reinforcement Therapy
- Standard treatment (Placebo Comparator): Standard treatment
  Interventions: Behavioral: Standard treatment

INTERVENTIONS:
Behavioral: Circadian Reinforcement Therapy — Circadian reinforcement therapy plus electronical monitoring. Circadian reinforcement therapy is a specialized psychoeducation working with strengthening of circadian rhythms.
  Arms: Circadian Reinforcement Therapy
Behavioral: Standard treatment — Standard treatment plus electronical monitoring
  Arms: Standard treatment

SUMMARY:
Very little is known of depressed patients' mental state after being discharged from inpatient wards where they are provided with a sheltered environment with stable sleep wake cycle, regular meals, and regular physical and social activities. Our previous usability study, SAFE I, showed that electronic self-monitoring was a useful tool to gain insight into patients' condition in the weeks after discharge. Results showed that patients over a four week period had significant day to day variations in self-rated mood and sleeping schedule and that the patients' sleep patterns were delayed with 45 minutes.

In the actual study, SAFE II, we are investigating whether an intervention with a strong focus on the circadian timing of daytime activities, and sleep, coined Circadian Reinforcement Therapy (CRT), can lead to a faster recovery of depression and prevent relapse into depression after discharge.

DETAILED DESCRIPTION:
SAFE II Background Patients hospitalized with a depression are generally discharged within 4-6 weeks, but remain vulnerable, and not fully recovered at discharge, hence a majority will be referred to outpatient care. Often, however, patients have to wait for about 2 weeks from discharge to first visit in the outpatient clinic. Our clinical experience is that this period from discharge to start of outpatient care is associated with psychological uncertainty and often cause unstable daily routines for sleep, meals, social life, and exercise. This may result in aggravation of the depression with the associated risk of suicidal thoughts and readmission. Our first study "E-monitoring by depression - Safe I," illustrated these issues. Patients registered their state daily in an electronical application, for sleep, mood, and exercise. Among other things the study showed that the patients' sleep patterns were advanced to later in the evening and longer in the morning thus shifting the sleep-wake cycle to later. One possible explanation for this finding is that patients are not recovered from the depression when discharged and therefore are more vulnerable to changes. Another possible factor is that at home the patients do not have the same support to keep daily structure as during hospitalization. This project "Safe discharge - SafeII" is based on the experience from the first study and will investigate whether a focused intervention in the benefits of a stable sleep in the recovery of a depression can help prevent worsening of the depression in the waiting time for outpatient treatment. It is well documented that stable sleep and circadian rhythm is an important element in the recovery of a depression.

Aim The purpose is to examine whether focused guidance to improve sleep habits and circadian rhythms can speed up recovery and also prevent worsening of depression and thus prevent readmission.

Design and Methods All patients hospitalized at PCK (Psychiatric Center Copenhagen) with a unipolar depression, and referred to outpatient treatment at the Intensive outpatient unit for affective disorders) (IAA) at discharge, are eligible for inclusion. Patient agreeing to participate will be randomized to one of two groups. The standard care group consists of patients who will be asked to register their mental state on a daily basis (mood, sleep and exercise) in the electronical application Daybuilder (www.Daybuilder.com). This standard group will have weekly telephone contact with the investigators. The intervention group will also be asked to register their daily state in the Daybuilder app and have weekly telephone contact with the investigators. In addition to standard care this group will also receive individual guidance concerning the importance of stabilization of the sleep-wake cycle and sleep to recover from depression. The primary outcomes of the study are changes in self-rated mood and changes in Hamilton depression rating scores at baseline and endpoint in the two groups and number of readmissions. We expect that the intervention group will have a more rapid recovery of depression and have fewer readmissions. Furthermore, in a subset of patients, the levels of the sleep hormone melatonin, a biological marker of circadian rhythms, is measured, as a profile to establish the dim light melatonin onset (DLMO) at the start and end of the intervention. At total of 150 patients, 75 in each group will be included in the project over a three year period In this study we get the opportunity to see the isolated impact of focusing on sleep and circadian rhythm in the recovery from depression. We have coined this intervention Circadian Reinforcement Therapy (CRT).

Implications If the findings are positive, we expect to implement the intervention more systematically in the psychiatric services thereby improving the conditions of patients with depression by making the transition from in- to outpatient status less risky and more stable. In the long term perspective the intervention can underpin recovery from depression, and prevent relapse into depression and readmission in mental hospital.

ELIGIBILITY:
Inclusion Criteria:

* Major depression as defined in DSM-5
* Hospitalized at a psychiatric inpatient ward
* Age above 18

Exclusion Criteria:

* Bipolar depression
* Suicidal plans or ideations (score of 2 or more on the HAM-D17 scale) item 3 or if investigator is unsure of level og suicidality
* Dementia or other organic brain damage that might influence ability to use the electronical monitoring system (Daybuilder) and the rules of the study
* Psychotic depression at time of inclusion.
* Abuse of alcohol or other drugs that might influence the ability to comply with study rules
* Patients under any form of coercion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Mood | 28 days
  Selfassessed mood rating from electronically entered data

SECONDARY OUTCOMES:
Readmission | 28 days
  Number of readmissions
Interviewer based mood | 28 days
  Hamilton depression rating scale scores

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatic Hospital Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The Danish National Archives

REFERENCES:
- [Derived] Aggestrup AS, Svendsen SD, Praestegaard A, Loventoft P, Norregaard L, Knorr U, Dam H, Frokjaer E, Danilenko K, Hageman I, Faurholt-Jepsen M, Kessing LV, Martiny K. Circadian Reinforcement Therapy in Combination With Electronic Self-Monitoring to Facilitate a Safe Postdischarge Period for Patients With Major Depression: Randomized Controlled Trial. JMIR Ment Health. 2023 Nov 27;10:e50072. doi: 10.2196/50072. PMID 37800194
- [Derived] Dunker Svendsen S, Aggestrup AS, Norregaard LB, Loventoft P, Praestegaard A, Danilenko KV, Frost M, Knorr U, Hageman I, Vedel Kessing L, Martiny K. Circadian reinforcement therapy in combination with electronic self-monitoring to facilitate a safe post-discharge period of patients with depression by stabilizing sleep: protocol of a randomized controlled trial. BMC Psychiatry. 2019 Apr 25;19(1):124. doi: 10.1186/s12888-019-2101-z. PMID 31023274